CLINICAL TRIAL: NCT04989751
Title: A Multicenter Phenotype-Genotype Analysis of Limb Girdle Muscular Dystrophy Patients in China
Brief Title: A Multicenter Phenotype-Genotype Analysis of LGMD Patients in China
Status: Enrolling by invitation | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Professor, Huashan Hospital
Other Study IDs: KY2019-409
Record Dates: First submitted 2021-08-02; First posted 2021-08-04 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: LGMD; LGMDR2; LGMDR1
Keywords: Observational
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2B; Limb-girdle muscular dystrophy type 2A | interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Muscle tissue was frozen with liquid nitrogen as soon as possible following excision and maintained at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMD patients
  Interventions: Diagnostic Test: Electromyography; Diagnostic Test: IDEAL MRI

INTERVENTIONS:
Diagnostic Test: Electromyography — Electromyography (EMG) would be used at the baseline for dignoisis and furtue analysis.
Diagnostic Test: IDEAL MRI — Muscle-speciifc sequences (e.g. IDEAL) would be used to scan patients at baseline and follow-up stages to characterize the fat fraction and atrophy in different muscles.

SUMMARY:
Limb-girdle muscular dystrophies (LGMD) are a series of rare progressive genetic disorders that are characterized by wasting and weakness of the voluntary proximal muscles. The onset of the disease is usually at young age, and most patients will be wheelchair-bound due to the progressive deterioration. Since currently genetic therapies for this disease are still immature, better natural history and genotype-phenotype studies are needed for preparing future therapies.

DETAILED DESCRIPTION:
This is multicentered-based, prospective, and observational study, which mainly focuses on the diagnosis and progression of limb-girdle muscular dystrophies (LGMD) in China. the investigators collect patient data including basic information, strength evaluations, genetic data, electromyography results, pathology imaging from muscle biopsies, and MRIs. Previously collected patient data may also be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Identified with variants regarding LGMD related genes revealed by genetic sequencing
* Progressive weakness involving shoulder girdle and/or pelvic girdle
* Myopathic changes in electromyography or in pathological studies

Exclusion Criteria:

* Identified with variants in other genes (non-LGMD related) that may cause muscular dystrophies

Min Age: 10 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The patients are mainly from neuromuscular diagnostic centers that participat this study in China.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in NSAA score | Baseline, Year 1, Year 3, Year 5
  The North Star Ambulatory Assessment (NSAA) is a 17-item rating scale with a score range of 0-34. It is used to measure the functional motor abilities of ambulant patients with muscular dystrophy. A lower NSAA score indicates more severe damage to the participant's motor capability.

SECONDARY OUTCOMES:
Changes in muscle fat infiltration | Baseline, Year 3, Year 5
  The muscle-specific fat fraction can be calculated with special MRI sequences such as IDEAL or Dixon in the region of interest. An deep-learning based tool is applied to segment individual muscles.
Changes in 6 Minute Walk Test | Baseline, Year 3, Year 5
  The 6-Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered in 6 minutes serves as the outcome for comparing changes in performance capacity.
Changes in 10 Metre Walk Test (10MWT) | Baseline, Year 3, Year 5
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, PhD, Study Director — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China